CLINICAL TRIAL: NCT02395835
Title: Methylation Evaluation of the PPARg Promoter Region (-351 to -260) in Pregnancy
Brief Title: Methylation of the PPARg Promoter Region in Pregnancy
Status: Completed | Type: Observational
Sponsor: Materno-Perinatal Hospital of the State of Mexico (Other)
Responsible Party: Principal Investigator, Hugo Mendieta Zeron, Médico Internista adscrito a la Unidad de Cuidados Intensivos Obstétricos, Materno-Perinatal Hospital of the State of Mexico
Other Study IDs: 05-06-2009
Record Dates: First submitted 2015-03-11; First posted 2015-03-24 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2015-03

CONDITIONS: Body Weight
Keywords: body mass index; methylation; PPAR gamma; pregnancy
MeSH Terms: conditions — Body Weight

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — Leukocytes were obtained according to the ACK-lysing buffer (LONZA) protocol. Briefly, a peripheral blood sample was placed in EDTA tube and then centrifuged at 2500 rpm for 10 min. All samples were kept at -80°C until further analysis.
  DNA was extracted from leukocytes (4000-10,000 cells) in the MagnaPure (Roche) using the MagNAPure LC DNA Isolation Kit 1 (Roche, Germany).
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Normal weight (NW) pregnant women: Pregnant women with Body Mass Index (BMI) > = 30. Body weight and height were measured in an overnight fasting status using an adult scale (Seca, Hamburg, Germany). Prepregnancy BMI was calculated as weight in kg divided by height in meters squared based on the prenatal chart or on the self-reported weight of women with no prenatal chart.
  Dietetic treatment was calculated according to height, weeks of gestation, and weight, considering an energy intake of 30 kcal/kg of ideal weight and a macronutrient distribution of: 55-65% carbohydrates, 10-20% fat, and the remainder as proteins.
- Overweight (OW) pregnant women: Pregnant women with Body Mass Index (BMI) < 30. Body weight and height were measured in an overnight fasting status using an adult scale (Seca, Hamburg, Germany). Prepregnancy BMI was calculated as weight in kg divided by height in meters squared based on the prenatal chart or on the self-reported weight of women with no prenatal chart.
  Dietetic treatment was calculated according to height, weeks of gestation, and weight, considering an energy intake of 30 kcal/kg of ideal weight and a macronutrient distribution of: 55-65% carbohydrates, 10-20% fat, and the remainder as proteins.

SUMMARY:
The main objective of this study was to assess whether clinical, anthropometric, and biochemical variables of the mother were associated with changes in the methylation of the PPARg promoter region (-351 to -260). Methodology: This was a matched cohort study with two groups: a) normal weight (NW) pregnant women (n = 21) and their offspring, and b) overweight (OW) pregnant women (n = 20) and their offspring. DNA was extracted from leukocytes (4000-10,000 cells) in the MagnaPure (Roche) using the MagNAPure LC DNA Isolation Kit 1 (Roche, Germany). The treatment of DNA (2 µg) was performed with sodium bisulfite (EZ DNA Methylation-Direct Kit, ZymoResearch). Real-time polymerase chain reaction (qPCR) was performed in a LightCycler 2.0 (Roche) using the SYBR® Advantage® qPCR Premix Kit (Clontech).

DETAILED DESCRIPTION:
Women were recruited in the first trimester of pregnancy not including cases with congenital heart and disabling or autoimmune diseases. Those whose clinical follow-up were lost or, if in the postpartum period, who had to be attended in the obstetric intensive care unit were eliminated from the study.

A clinical visit per month was established. Body weight and height were measured in an overnight fasting status using an adult scale (Seca, Hamburg, Germany). Prepregnancy Body Mass Index (BMI) was calculated as weight in kg divided by height in meters squared based on the prenatal chart or on the self-reported weight of women with no prenatal chart.

Blood pressure was recorded at each visit using a standard sphygmomanometer (Riester Big Ben® Square, Germany). Preeclampsia was diagnosed and classified according to the American College of Obstetricians and Gynecologists (ACOG).

Fasting blood samples (10 ml) were taken at the HMPMP laboratory in an early morning after an overnight fasting. Serum samples were analyzed for glucose and lipid profile (Dimension Rx L Max, Dade Behring, USA). At the end of pregnancy, 1 to 2 ml of neonatal peripheral blood sample for leukocyte DNA extraction was taken.

Dietetic treatment was calculated according to height, weeks of gestation, and weight, considering an energy intake of 30 kcal/kg of ideal weight and a macronutrient distribution of: 55-65% carbohydrates, 10-20% fat, and the remainder as proteins. On each nutritional visit, the Healthy Eating Index for Pregnancy (HEI) was evaluated, and all women were recommended to include methionine-rich foods (beans, eggs, fish, garlic, lentils, onion, and soy) and those containing folic acid and vitamin B12 (beef liver, cereals, whole grains, yeast, etc.) in adequate quantities in their diet. The information was complemented with the Food Frequency Questionnaire (FFQ), and the diet adherence was considered adequate with 80% compliance to the indicated calories, at least in four visits.

This project had no risk to pregnant women and their infants, according to the regulations of the General Health Research Law of Mexico. We followed the Declaration of Helsinki, and all patients were asked to sign the written informed consent.

ELIGIBILITY:
Inclusion Criteria: Women attended in the first trimester of pregnancy -

Exclusion Criteria: congenital heart and disabling or autoimmune diseases

-

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant women attended at the Maternal-Perinatal Hospital "Mónica Pretelini Sáenz".
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2009-09; Primary Completion 2010-08 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Evidence of the effect of Body Mass Index (BMI) on the methylation status of the PPAR gamma promoter region (-351 to -260). | Pregnant women were followed until delivery.
  The treatment of DNA (2 µg) was performed with sodium bisulfite (EZ DNA Methylation-Direct Kit, ZymoResearch). For the control group, we used purified human methylated and unmethylated DNA (Zymo Research) with specific oligonucleotides. Lymphocyte DNA from healthy donors was used as negative control, and methylated DNA "in vitro" with Sss I enzyme (New England Biolabs) was used as positive control for methylation.
  The methylated (M3) and unmethylated (U3) primers used were those proposed by Pancione et al.

CONTACTS AND LOCATIONS:
Overall Officials: Hugo Mendieta Zerón, PhD., Principal Investigator — Asociación Científica Latina A.C.